CLINICAL TRIAL: NCT04396145
Title: The Effects of Chronic Otitis Surgery on Virtual Subjective Vertical
Brief Title: The Effects of Chronic Otitis Surgery on SVV
Status: Active, not recruiting | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Fazıl Necdet Ardıç, Chief Department of Otolaryngology, Pamukkale University
Other Study IDs: 5
Record Dates: First submitted 2020-05-17; First posted 2020-05-20 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Chronic Otitis Media

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Surgery group: Subjects who will have chronic otitis media surgery will be included in the study.
  Interventions: Diagnostic Test: Subjective Visual Vertical

INTERVENTIONS:
Diagnostic Test: Subjective Visual Vertical — All subjects will have Virtual SVV before and after the operation

SUMMARY:
Inner ear trauma during chronic otitis surgery is one of the major concerns of Otolaryngology. Hearing thresholds or semicircular canals were investigated with this purpose. The investigator's aim is to test the utricle for surgical trauma.

DETAILED DESCRIPTION:
All patients who will have surgery for ear will be tested before the operation and after the first day and the first week. Virtual SVV(Interacoustics) will be used for testing. The deviation angle from the vertical line will be measured when 15, 30, and 45-degree head tilt to the left and right side while they were standing.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Otitis Media
* Who had surgical treatment

Exclusion Criteria:

* A patient who had the vestibular disease before
* Neurologic disease
* Patients who had ear, brain and musculoskeletal surgery before

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic otitis media
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-04-29 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
SVV angle | 1 week
  Right and Left deviation angle when head tilted 15, 30, and 45 degree

CONTACTS AND LOCATIONS:
Overall Officials: Fazıl N Ardıç, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data will be available in university depository